CLINICAL TRIAL: NCT06075277
Title: Relative Bioavailability of BI 1810631 Following Oral Administration Under Fed and Fasted Conditions in Healthy Male Subjects (an Open-label, Randomised, Single-dose, Two-way Crossover Trial)
Brief Title: A Study in Healthy Men to Test How Zongertinib is Taken up in the Body When Taken With or Without Food
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1479-0010; 2022-502860-19-00 (Registry Identifier: CTIS (EU)); U1111-1291-3312 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2023-10-04; First posted 2023-10-10 (Actual); Results first posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: two-way crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- BI 1810631 (iCF) fed state (Reference, R) then fasting state (Test, T) (Experimental): Period 1: Participants received a single oral dose of 240 milligram (mg) Zongertinib as film coated tablets (4x 60 mg tablet) following a high fat/high calorie meal.
  Period 2: Participants received a single oral dose of 240 milligram (mg) of Zongertinib as film coated tablets (4x 60 mg tablets) following an overnight fast of at least 10 hours.
  Interventions: Drug: zongertinib
- BI 1810631 (iCF) fasting state (Test, T) then fed state (Reference, R) (Experimental): Period 1: Participants received a single oral dose of 240 milligram (mg) of Zongertinib as film coated tablets (4x 60 mg tablets) following an overnight fast of at least 10 hours.
  Period 2: Participants received a single oral dose of 240 milligram (mg) Zongertinib as film coated tablets (4x 60 mg tablet) following a high fat/high calorie meal.
  Interventions: Drug: zongertinib

INTERVENTIONS:
Drug: zongertinib — Participants received a single oral dose of 240 mg Zongertinib (4 x 60 mg tablets) in two periods: in Period 1 after an overnight fast of at least 10 hours, and in Period 2 following a high fat/high calorie meal.
  Other Names: BI 1810631, Hernexeos®

SUMMARY:
The main objective of this trial is to investigate the relative bioavailability of a single dose of BI 1810631 intended commercial formulation (iCF) under fed (Test treatment, T) and fasted (Reference treatment, R) conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
2. Age of 18 to 55 years (inclusive)
3. Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
4. Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial

Exclusion Criteria:

1. Any finding in the medical examination (including Blood pressure (BP), pulse rate (PR) or electrocardiogram (ECG)) deviating from normal and assessed as clinically relevant by the investigator
2. Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
4. Any evidence of a concomitant disease assessed as clinically relevant by the investigator
5. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
6. Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
7. Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
8. History of relevant orthostatic hypotension, fainting spells, or blackouts Further exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2023-10-19 (Actual); Primary Completion 2024-01-02 (Actual); Study Completion 2024-01-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Berlin GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label, randomized, two-way crossover design trial. Healthy males received a single oral dose of 240 mg Zongertinib (BI 1810631) in its intended commercial formulation (iCF) following an overnight fast and after a standardized high-calorie, high-fat meal. There was a washout period of 14 days between doses. The primary objective was to evaluate how Zongertinib is absorbed when taken with and without food, to determine differences in its bioavailability between these states.
Pre-assignment Details: All participants were screened for eligibility prior to participation in the trial. Participants attended a specialist site which ensured that they (the participants) strictly met all inclusion and none of the exclusion criteria. Participants were not to be allocated to a treatment sequence if any of the entry criteria were violated.
Groups:
- Zongertinib iCF Fasted (Reference (R)) /Zongertinib iCF Fed (Test (T)): Two period crossover separated by a wash-out of at least 14 days:
  Period 1: Participants received a single oral dose of 240 milligram (mg) of Zongertinib as film coated tablets (4x 60 mg tablets) following an overnight fast of at least 10 hours.
  Period 2: Participants received a single oral dose of 240 milligram (mg) Zongertinib as film coated tablets (4x 60 mg tablet) following a high fat/high calorie meal.
- Zongertinib iCF Fed (Test (T)) / Zongertinib iCF Fasted (Reference (R)): Two period crossover separated by a wash-out of at least 14 days:
  Period 1: Participants received a single oral dose of 240 milligram (mg) Zongertinib as film coated tablets (4x 60 mg tablet) following a high fat/high calorie meal.
  Period 2: Participants received a single oral dose of 240 milligram (mg) of Zongertinib as film coated tablets (4x 60 mg tablets) following an overnight fast of at least 10 hours.
Period: Period 1
Arm/Group | Zongertinib iCF Fasted (Reference (R)) /Zongertinib iCF Fed (Test (T)) | Zongertinib iCF Fed (Test (T)) / Zongertinib iCF Fasted (Reference (R))
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Washout Period
Arm/Group | Zongertinib iCF Fasted (Reference (R)) /Zongertinib iCF Fed (Test (T)) | Zongertinib iCF Fed (Test (T)) / Zongertinib iCF Fasted (Reference (R))
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Zongertinib iCF Fasted (Reference (R)) /Zongertinib iCF Fed (Test (T)) | Zongertinib iCF Fed (Test (T)) / Zongertinib iCF Fasted (Reference (R))
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The treated set includes all subjects who were treated with at least one dose of trial drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Zongertinib iCF Fasted (Reference (R)) /Zongertinib iCF Fed (Test (T)) | Zongertinib iCF Fed (Test (T)) / Zongertinib iCF Fasted (Reference (R)) | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.0 (5.8) | 45.9 (11.2) | 47.9 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 8 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 8 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 8 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of Zongertinib in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of Zongertinib in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz).
  Geometric least square mean (adjusted geometric mean) and geometric standard error were calculated using an analysis of variance (ANOVA) model on the logarithmic scale. The pharmacokinetic (PK) endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model. These quantities will then be back-transformed to the original scale to provide the point estimate and 90% confidence intervals (CIs) for each endpoint.
Time Frame: Within 3 hours before Zongertinib administration, and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144, and 168 hours following administration.
Population: Pharmacokinetic parameter analysis set (PKS): all subjects who were randomised and received at least one dose of trial medication and who provided at least one pharmacokinetic (PK) endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability.
Measure: Geometric Mean (Standard Error); unit: hour*nanomol/Liter (h*nmol/L)
Groups:
- Zongertinib iCF Fed (Test (T)): Participants received a single oral dose of 240 milligrams (mg) of Zongertinib as film-coated tablets (4 x 60 mg tablets) following a high-fat, high-calorie meal.
- Zongertinib iCF Fasted (Reference (R)): Participants received a single oral dose of 240 milligrams (mg) of Zongertinib as film-coated tablets (4 x 60 mg tablets) following an overnight fast of at least 10 hours.
Arm/Group | Zongertinib iCF Fed (Test (T)) | Zongertinib iCF Fasted (Reference (R))
Number analyzed (Participants) | 16 | 16
hour*nanomol/Liter (h*nmol/L) | 59457.92 (NA) — Geometric standard error = 1.07 | 46951.21 (NA) — Geometric standard error = 1.07
Statistical Analysis 1: Comparison: Zongertinib iCF Fed (Test (T)) vs Zongertinib iCF Fasted (Reference (R)); Relative bioavailability of Zongertinib administered in fed state (Test) compared with Zongertinib administered in fasted state (Reference) was estimated by the ratios of the gMeans (Test/Reference). Their corresponding 2-sided 90% confidence intervals (CIs) were provided. This method corresponds to 2 one-sided t-test procedures, each at the 5% significance level; Test type: Other; Ratios of adjusted geometric means [%] = 126.64, 90% CI 2-sided [112.09 to 143.08] — Ratio calculated as test/reference*100. Intra-individual Geometric coefficient of variation [%] = 19.8

2. Primary Outcome: Maximum Measured Concentration of the Zongertinib in Plasma (Cmax)
Description: Maximum measured concentration of Zongertinib in plasma (Cmax).
  Geometric least square mean (adjusted geometric mean) and geometric standard error were calculated using an analysis of variance (ANOVA) model on the logarithmic scale. The pharmacokinetic (PK) endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model. These quantities will then be back-transformed to the original scale to provide the point estimate and 90% confidence intervals (CIs) for each endpoint.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: nanomol/Liter (nmol/L)
Arm/Group | Zongertinib iCF Fed (Test (T)) | Zongertinib iCF Fasted (Reference (R))
Number analyzed (Participants) | 16 | 16
nanomol/Liter (nmol/L) | 4666.87 (NA) — Geometric standard error = 1.09 | 3700.37 (NA) — Geometric standard error = 1.09
Statistical Analysis 1: Comparison: Zongertinib iCF Fed (Test (T)) vs Zongertinib iCF Fasted (Reference (R)); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratios of adjusted geometric means [%] = 126.12, 90% CI 2-sided [106.34 to 149.58] — Ratio calculated as test/reference*100. Intra-individual Geometric coefficient of variation [%] = 27.9

3. Secondary Outcome: Area Under the Concentration-time Curve of Zongertinib in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of Zongertinib in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞).
  Geometric least square mean (adjusted geometric mean) and geometric standard error were calculated using an analysis of variance (ANOVA) model on the logarithmic scale. The pharmacokinetic (PK) endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model. These quantities will then be back-transformed to the original scale to provide the point estimate and 90% confidence intervals (CIs) for each endpoint.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: hour*nanomol/Liter (h*nmol/L)
Arm/Group | Zongertinib iCF Fed (Test (T)) | Zongertinib iCF Fasted (Reference (R))
Number analyzed (Participants) | 16 | 16
hour*nanomol/Liter (h*nmol/L) | 59986.25 (NA) — Geometric standard error = 1.07 | 47594.57 (NA) — Geometric standard error = 1.07
Statistical Analysis 1: Comparison: Zongertinib iCF Fed (Test (T)) vs Zongertinib iCF Fasted (Reference (R)); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratios of adjusted geometric means [%] = 126.04, 90% CI 2-sided [111.70 to 142.21] — Ratio calculated as test/reference*100. Intra-individual Geometric coefficient of variation [%] = 19.6

ADVERSE EVENTS:
Time Frame: Serious Adverse Events and other adverse events: From first Zongertnib dose up to 14 days. All-cause mortality: From first trial drug administration up to 22 days
Description: Population description: Treated set (TS)- The treated set includes all subjects who were treated with at least one dose of trial drug.
Groups:
- Zongertinib 240mg iCF Fed (T): Participants received a single oral dose of 240 milligrams (mg) of Zongertinib as film-coated tablets (4 x 60 mg tablets) following a high-fat, high-calorie meal.
- Zongertinib 240mg iCF Fast (R): Participants received a single oral dose of 240 milligrams (mg) of Zongertinib as film-coated tablets (4 x 60 mg tablets) following an overnight fast of at least 10 hours.
Arm/Group | Zongertinib 240mg iCF Fed (T) | Zongertinib 240mg iCF Fast (R)
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 7/16 | 7/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zongertinib 240mg iCF Fed (T) (N=16) | Zongertinib 240mg iCF Fast (R) (N=16)
Nausea (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 3
Presyncope (Nervous system disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-11-13): https://cdn.clinicaltrials.gov/large-docs/77/NCT06075277/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-15): https://cdn.clinicaltrials.gov/large-docs/77/NCT06075277/SAP_001.pdf